CLINICAL TRIAL: NCT02379013
Title: Development and Evaluation of a Cognitive-motor System for a Quantitative and Objective Measure of Fatigue in Functional MRI
Brief Title: Measure of Fatigue in Functional MRI
Acronym: FATIGUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Collaborators: Paris West University Nanterre La Défense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRD0714
Record Dates: First submitted 2015-01-26; First posted 2015-03-04 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Fatigue
Keywords: Fatigue; functional MRI
MeSH Terms: conditions — Fatigue | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volunteer with MRI (Experimental): All volunteer will be included in the arm MRI
  Interventions: Procedure: Volunteer with MRI

INTERVENTIONS:
Procedure: Volunteer with MRI — functional MRI

SUMMARY:
The purpose of this study is to determine more objective, central and peripheral indices of fatigue state by exploring the neural and behavioral correlates of the alert process while keeping the idea to corroborate these results with those obtained during the performance of physical exercises and neuropsychological tests "classics" of attention, motivation, and functions evaluation. The interest of this study is to manipulate and compare the phasic and tonic alert mechanism through the activation of an extrinsic motivational system during fatigue. The investigators have chosen the alert since it is a basic cognitive process defined as the ability to increase attentional resources with the expectation of a target stimulus resulting in reduced response time. It can be phasic (extrinsic), favored by the presence of a warning signal preceding the target (preparation time) or tonic (intrinsic) occurring without warning signal (wakefulness). The evaluation of the alert is classically realized by a simple reaction time task with the presence or not of warning signal soliciting wether the tonic alert or the phasic alert.

The investigators suppose to revisit the healthy population with brain model alert issued in 2010 which highlighted the predominant role of the regions of the dorsolateral prefrontal cortex, parietal, cingulate and thalamus (non-motor) in maintaining attention and temporal preparation alert task.

The investigators identify also functional, motor and cognitive components of basal ganglia of thalamus. Cognitive-motor paradigm and neurological dysfunctions observed in multiple sclerosis population will help to identify and separate the cognitive role and motor brain regions, particularly the thalamus and basal ganglia. New neurological hypotheses are proposed

DETAILED DESCRIPTION:
This project will be applied on healthy subjects, and the subject will be equipped with two electrodes attached to the muscle of the left arm (flexor) to measure muscle activity. That will be performed with a handgrip (the subject press on the handgrip).The subject will receive two sessions. It will conduct a trial session in the laboratory to control his ability to imagine the task (imagination run) and perform the driving task correctly.

Two saliva samples will be placed in tubes to be analysed to measure the concentration of cortisol before and after functional MRI. Then, psychological and satisfaction questionnaires will be completed by volunteers.

This protocol will then be adapted and transferred to multiple sclerosis population (in a second study), for which fatigue is one of the symptoms most commonly reported.

ELIGIBILITY:
Inclusion Criteria:

* Male or female right-handed aged between 18 and 35 years
* Free of neurological, psychiatric or abuse of alcohol or drugs
* Affiliated with the social security system (beneficiary or legal)
* Having understood the information and having signed the consent form

Exclusion Criteria:

* Against indication to 'MRI': Pacemaker or neurosensory pacemaker or implantable defibrillator, cochlear implants, Ocular or cerebral ferromagnetic foreign body near the nerve structures, metal prosthesis, Ventriculoperitoneal shunt valves neurosurgical, brace, Agitation of the patient: not cooperating or agitated subjects, low-age children, claustrophobic patient, expectant mother
* Front-temporal dementia
* Physical or psychiatric illness likely to interfere with the functional assessment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assessment of executive function and circuit of functional MRI | 1 day
  Brain activity will be measured during tests to determine the central indices and peripheral quantitative and objectives of the state of fatigue.

SECONDARY OUTCOMES:
Muscle strength measured with the electromyogram data | 1 day
  This outcome will be measured with the electromyogram data
Saliva samples to measure the concentration of cortisol | 1 day
  Samples will be placed in tubes to be analysed to measure the concentration of cortisol.
Assess attentional and executive functions (questionnaires) | 1 day
  Results of psychological (Mesulam, D2, Stroop) questionnaires
Evaluation of voluntary satisfaction (questionnaire) | 1 day
  satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alain LE BLANCHE, PUPH, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No